CLINICAL TRIAL: NCT06930989
Title: Twin Threat of OSA and Hypertension on Mortality/CV-risk and Protective Effect by Positive Airway Pressure Treatment.
Brief Title: Primary Prevention Long-term Registry Study in OSA and Hypertension. Survival Analysis 2010-2022
Acronym: DISCOVERY-HT
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Swedish Heart Lung Foundation (Other); Göteborg University (Other); Lund University (Other); Uppsala University (Other)
Responsible Party: Principal Investigator, Sven Svedmyr, MD, principal investigator, Vastra Gotaland Region
Other Study IDs: SERA Lund DNR:2025-00712-02
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; OSA - Obstructive Sleep Apnea; MACE; Survival Analysis; PAP
Keywords: Primary CV prevention; hypertension; OSA; PAP
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hypertension and obstructive sleep apnea (OSA): Patients with hypertension and positive airway pressure (PAP) treated OSA
  Interventions: Device: Positive airway pressure (PAP)
- OSA alone: Patients with PAP teated OSA but no hypertension
  Interventions: Device: Positive airway pressure (PAP)
- Hypertension control: Patients of control population with hypertension
- Healthy controls: Control population without hypertension and without OSA

INTERVENTIONS:
Device: Positive airway pressure (PAP) — Intervention as part of routine clinical care. Data from national registries.
  Groups: Hypertension and obstructive sleep apnea (OSA); OSA alone

SUMMARY:
Hypertension and obstructive sleep apnea (OSA) are both common conditions that independently increase the risk cardiovascular disease including atrial fibrillation, ischemic heart disease, heart failure and stroke. OSA is also an independent promoter of hypertension development and poorly controlled hypertension is overrepresented in OSA. Finally, HT and OSA share many risk factors including obesity, and several lifestyle factors. Altogether, these links contribute to a high prevalence of patients with both disorders.

The investigators suspect participants with HT and OSA are at even higher CV risk and may get their first CV event earlier in life. Comparison between HT and OSA participants vs HT alone, OSA alone or healthy controls has not previously been investigated in large studies.

Thus, the investigators aim to investigate long-term risk of major cardiovascular events (MACE) or death comparing these groups in registry data between 2010-2022 in Sweden. The investigators will also investigate the protecting effect of positive airway pressure (PAP) on the OSA related CV risk increase and how many hours/night of PAP use is needed to get any protective effects.

DETAILED DESCRIPTION:
Please see attached analysis plan

ELIGIBILITY:
Inclusion Criteria:

* Adult patients starting PAP treatment for OSA in the swedevox registry between 2010-2021 with and without hypertension. Randomly selected controls with and without hypertension from the general population.

Exclusion Criteria:

* Patients with manifest cardiovascular disease (stroke, ischemic heart disease, cardiac failure or atrial fibrillation at baseline).
* Patients with kidney failure at baseline.
* Patients with malignant cancer at baseline.
* Subjects with missing data on any of the main variables in the fitted models.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Discovery ("Course of DISease in patients reported to the Swedish CPAP Oxygen and VEntilator RegistrY") 2.0 is a large clinical cohort on patients with home mechanical ventilation, long-term oxygen treatment and/or CPAP treatment with data from the Swedish national register for patients on Long Term Oxygen Therapy and Home Mechanical Ventilation (Swedevox) and the Swedish Sleep Apnea Registry (SESAR). Data are cross referenced using Swedish personal IDs with data from multiple Swedish national registries including the National Patients diagnosis registry, National prescription registry, National Cause of Death Register, and SCBs registries on socioeconomic information. All patients starting PAP treatment for OSA during 2010-2021 are included.
Sampling Method: Probability Sample
Enrollment: 148467 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Major cardiovascular event (MACE) | First event during follow-up 2010-2022
  Major cardiovascular event (MACE) including CV death
Age at first MACE | First event during follow-up 2010-2022
  mean age at first MACE for the groups
All cause death | 2010-2022
  death from any cause during follow-up

SECONDARY OUTCOMES:
Risk reduction with PAP | 2010-2022
  Survival analysis between both OSA groups only stratified by PAP adherence (hours/night)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Svedmyr, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital and Göteborg University, Gothenburg, VGR, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data can be made available from the discovery cohort on case to case basis after applying to the discovery cohort registry holder after reasonable request.
Supporting Information: SAP
Time Frame: SAP will be public here. Original data is property of the Discovery registry, see above.
Access Criteria: SAP here. Data see above.

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT06930989/SAP_001.pdf